CLINICAL TRIAL: NCT05345873
Title: A Randomized, Double-blind, Positive-controlled Phase II Clinical Trial to Evaluate the Immunogenicity and Safety of SCTV01E (A COVID-19 Alpha/Beta/Delta/Omicron Variants S-Trimer Vaccine) in Adolescents Aged 12-17 Years and Previously Fully Vaccinated With mRNA COVID-19 Vaccine
Brief Title: A Study to Evaluate the Immunogenicity and Safety of a Recombinant Protein COVID-19 Vaccine as a Booster Dose in Population Aged 12-17 Years
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sinocelltech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SCTV01E-01-mRNA-THA-1
Record Dates: First submitted 2022-04-25; First posted 2022-04-26 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: COVID-19; SARS-CoV-2 Infection
Keywords: COVID-19; SARS-CoV-2; Vaccine
MeSH Terms: conditions — COVID-19 | interventions — SCTV01C vaccine; 2019-nCoV Vaccine mRNA-1273

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SCTV01E Group (Experimental): one dose of SCTV01E, intramuscular
  Interventions: Biological: SCTV01E
- mRNA-1273 (Active Comparator): one dose of mRNA-1273, intramuscular
  Interventions: Biological: mRNA-1273

INTERVENTIONS:
Biological: SCTV01E — one dose of SCTV01E on D0, intramuscular
  Arms: SCTV01E Group
Biological: mRNA-1273 — one dose of mRNA-1273 on D0, intramuscular
  Arms: mRNA-1273

SUMMARY:
The study is a randomized, double-blind, positive-controlled Phase II booster study. It will evaluate the immunogenicity and safety of SCTV01E compared with mRNA-1273 (the mRNA COVID-19 vaccine from Moderna) in population aged 12-17 years old and previously vaccinated with 2 doses of mRNA COVID-19 vaccine.

DETAILED DESCRIPTION:
Approximately 300 participants aged 12-17 years old and previously vaccinated with 2 doses of mRNA COVID-19 vaccine (Comirnaty from Pfizer or mRNA-1273 from Moderna, participants previously vaccinated with mRNA1273 are more preferred) will be enrolled in this study and be randomly assigned to SCTV01E Group and mRNA-1273 Group in a ratio of 1:1.

ELIGIBILITY:
Inclusion Criteria:

* Participants are eligible to be included in the study only if the following conditions are met:

  1. Male or female aged 12-17 years old when signing ICF;
  2. Participants who were fully vaccinated with 2 doses of mRNA COVID-19 vaccine (mRNA-1273 from Moderna or Comirnaty from Pfizer, participants previously vaccinated with mRNA1273 are more preferred) and the interval between the last dose and this study vaccination is 3 to 12 months;
  3. The participant and/or his legal guardian can sign written ICF, and can fully understand the trial procedure, the risk of participating in the trial, and other interventions that can be selected if they do not participate in the trial;
  4. The participant and/or his legal guardian has the ability to read, understand, and fill in record cards;
  5. Healthy participants or participants with pre-existing medical conditions who are in stable condition. The "pre-existing medical conditions" include but not limited to hypertension, diabetes, chronic cholecystitis and cholelithiasis, chronic gastritis that meet the described criteria. A stable medical condition is defined as disease not requiring significant change in therapy or no need for hospitalization as a consequence of worsening disease state for at least 3 months prior to enrollment;
  6. Fertile men and women of childbearing potential voluntarily agree to take effective contraceptive measures from signing ICF to 6 months after the study vaccination; the pregnancy test results of women of childbearing potential are negative on screening.

Exclusion Criteria:

* A participant who conforms to any of the following criteria should be excluded from the study:

  1. Presence of fever within 3 days before the study vaccination;
  2. A positive result of nucleic acid test for SARS-CoV-2 during the screening period or previously diagnosed with COVID-19;
  3. A history of infection or disease related to severe acute respiratory syndrome (SARS), Middle East respiratory syndrome (MERS), or other disease with corresponding use of immunosuppressants;
  4. A history of allergic reactions to any vaccine or drug, such as allergy, urticaria, severe skin eczema, dyspnea, laryngeal edema, and angioneurotic edema;
  5. A medical or family history of seizure, epilepsy, encephalopathy and psychosis;
  6. Immunocompromised patients suffering from immunodeficiency diseases, important organ diseases, immune diseases (including Guillain-Barre Syndrome [GBS], systemic lupus erythematosus, rheumatoid arthritis, asplenia or splenectomy caused by any circumstances, and other immune diseases that may have an impact on immune response in the investigator's opinion), etc.;
  7. Long-term use of immunosuppressant therapy or immunomodulatory drugs for ≥14 days within the first six months prior to enrollment. Whereas short-term (≤14 days) use of oral, inhaled and topical steroids are allowed;
  8. Patients on antituberculosis therapy;
  9. Presence of severe or uncontrollable cardiovascular diseases, or severe or uncontrollable disorders related to endocrine system, blood and lymphatic system, liver and kidney, respiratory system, metabolic and skeletal systems, or malignancies (skin basal cell carcinoma and carcinoma in-situ of cervix are exceptions and will not be excluded), such as severe heart failure, severe pulmonary heart disease, unstable angina, liver failure, or uremia;
  10. Contraindications for intramuscular injection or intravenous blood sampling, including thrombocytopenia and other blood coagulation disorders;
  11. Participants who received any immunoglobulin or blood products in the previous 3 months before enrollment, or plan to receive similar products during the study;
  12. Participants who received other investigational drugs within 1 month before the study vaccination;
  13. Participants who is at the acute stage of illness, such as acute onset of chronic heart failure, acute sore throat, hypertensive encephalopathy, acute pneumonia, acute renal insufficiency, acute cholecystitis;
  14. Participants received other drugs or vaccines used to prevent COVID-19, but participants previously received Vaxzevria will not be excluded;
  15. Participants vaccinated with influenza vaccine within 14 days or with other vaccines within 28 days before the study vaccination;
  16. Those who donated blood or had blood loss (≥450 mL) within 3 months before the vaccination or plan to donate blood during the study period;
  17. Those who are pregnant or breast-feeding or plan to be pregnant during the study period;
  18. Those who plan to donate ovum or sperms during the study period;
  19. Those who cannot follow the trial procedures, or cannot cooperate to complete the study due to planned relocation or long-term outing;
  20. Those unsuitable for participating in the clinical trial as determined by the investigator because of other abnormalities that are likely to confuse the study results, or non-conformance with the maximal benefits of the participants;
  21. Those who are tested positive for HIV.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2022-10-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Geometric mean titers (GMT) of neutralizing antibodies (nAb) to Omicron variant on Day 28 | Day 28 after the study vaccination
GMT of nAb to Delta variant on Day 28 | Day 28 after the study vaccination

SECONDARY OUTCOMES:
Number of IFN-γ positive (characterizing Th1) and IL-4 positive (characterizing Th2) T cell subsets on Day 28 | Day 28 after the study vaccination
Seroresponse rates of nAb to Omicron variant on Day 28 | Day 28 after the study vaccination
Seroresponse rates of nAb to Delta variant on Day 28 | Day 28 after the study vaccination
  Seroresponse is defined as a change of nAb from below the low limit of quantitation [LLOQ] to equal to or above LLOQ, or a ≥4-fold rise if baseline is equal to or above LLOQ in nAb from D0
Incidence and severity of solicited AEs from Day 0 to Day 7 after the study vaccination | Day 0 to Day 7 after the study vaccination
Incidence and severity of unsolicited AEs from Day 0 to Day 28 after the study vaccination | Day 0 to Day 28 after the study vaccination
Incidence and severity of SAEs and AESIs within 180 days after study vaccination | Day 0 to Day 180 after the study vaccination